CLINICAL TRIAL: NCT03486834
Title: Double-Blind, Randomized, Placebo-Controlled Phase 2b, Multi-center Study to Evaluate the Safety, Tolerability, Efficacy and Immunogenicity of a 2-Dose and a 3-Dose Regimen of V160 (Cytomegalovirus [CMV] Vaccine) in Healthy Seronegative Women, 16 to 35 Years of Age
Brief Title: V160 2-Dose and 3-Dose Regimens in Healthy Cytomegalovirus (CMV) Seronegative Females (V160-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V160-002; 2017-004233-86 (EudraCT Number)
Record Dates: First submitted 2018-03-28; First posted 2018-04-03 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Cytomegalovirus (CMV) Infections
Keywords: Prevention of cytomegalovirus infection (CMVi)
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- V160 3-Dose Regimen (Experimental): Participants received 3 doses of vaccine V160 (100 Units/0.5 mL dose with Merck aluminum phosphate adjuvant [MAPA], 4°C stable formulation) administered by intramuscular (IM) injection on Day 1, Month 2, and Month 6.
  Interventions: Biological: V160
- V160 2-Dose Regimen (Experimental): Participants received 2 doses of vaccine V160 (100 Units/0.5 mL dose with MAPA, 4°C stable formulation) administered IM on Day 1 and Month 6 and a placebo-saline solution at Month 2.
  Interventions: Biological: V160; Drug: Placebo
- Placebo (Placebo Comparator): Participants received placebo (saline solution) by IM injection on Day 1, Month 2, and Month 6.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: V160 — V160 was administered as a 0.5 mL (100 Units/0.5 mL dose with Merck aluminum phosphate adjuvant [MAPA], 4°C stable formulation) IM injection.
  Other Names: Human cytomegalovirus vaccine
  Arms: V160 2-Dose Regimen; V160 3-Dose Regimen
Drug: Placebo — Saline solution administered as a 0.5 mL IM injection
  Arms: Placebo; V160 2-Dose Regimen

SUMMARY:
This study evaluated the safety, tolerability, and efficacy of the cytomegalovirus (CMV) vaccine (V160) administered in a 2-dose or 3-dose regimen to healthy seronegative women 16 to 35 years of age. Participants received blinded V160 on Day 1, Month 2, and Month 6 (3-dose regimen), V160 on Day 1 and Month 6 and placebo at Month 2 (2-dose regimen), or placebo on Day 1, Month 2, and Month 6, and were followed to approximately Month 24. The primary hypothesis of the study was that administration of a 3-dose regimen of V160 will reduce the incidence of primary CMV infection compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy based on medical history and physical examination.
* Serologically confirmed to be CMV seronegative prior to receiving the first dose of V160/placebo
* Have direct exposure to young children (≤5 years of age) at home or occupationally
* Of childbearing potential
* Agrees to avoid becoming pregnant during the 6-month treatment period and for at least 4 weeks after the last dose of study drug by either 1) practicing abstinence from heterosexual activity, or 2) use a highly-effective method of birth control (as specified in the protocol) during heterosexual activity.

Exclusion Criteria:

* Has a history or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might expose the participant to risk by participating in the trial, confound the results of the trial, or interfere with participation for the full duration of the trial, as assessed by the investigator
* Has history of allergic reaction or anaphylactic reaction to any vaccine component that required medical intervention or of any severe allergic reaction to any vaccine component that required medical intervention.
* Has a recent (<72 hours) history of febrile illness (temperature ≥100.4°F/38.0°C, oral equivalent)
* Is currently immunocompromised or has been diagnosed as having a congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition that requires immunosuppressive medication.
* Has a condition in which repeated venipuncture or injections pose more than minimal risk for the participant.
* A woman of childbearing potential (WOCBP) who has a positive pregnancy test at screening or within 24 hours before the first dose of study treatment.
* Has previously received a CMV vaccine.
* Had any live virus vaccine administered or scheduled to be administered in the period from 4 weeks prior to, and 4 weeks following receipt of any dose of trial vaccine.
* Had any inactivated vaccine administered or scheduled within the period from 14 days prior to, through 14 days following, any dose of trial vaccine.
* Had administration of any immune globulin or blood product within 90 days prior to injection with V160/placebo or scheduled within 30 days thereafter.
* Received systemic corticosteroids (equivalent of ≥2 mg/kg total daily dose of prednisone or ≥20 mg/d for persons weighing >10 kg) for ≥14 consecutive days and has not completed treatment at least 30 days prior to trial entry.
* Received systemic corticosteroids exceeding physiologic replacement doses (≈5 mg/d prednisone equivalent) within 14 days prior to the first vaccination (participants using inhaled, nasal, or topical steroids are considered eligible for the trial).
* Received any anti-viral agent with proven or potential activity against CMV two weeks prior to vaccination or is likely to receive such an agent within 2 weeks after vaccination.
* Receiving or has received in the year prior to enrollment immunosuppressive therapies or other therapies used for solid organ/cell transplant, radiation therapy, immunosuppressive/cytotoxic immunotherapy, chemotherapy and other immunosuppressive therapies known to interfere with the immune response. Topical tacrolimus is allowed provided that it is not used within 2 weeks prior to, or 2 weeks following a V160 dose.
* Participated in another clinical trial in the past 4 weeks, or plans to participate in a treatment-based trial or a trial in which an invasive procedure is to be performed while enrolled in this trial.
* Plans donation of eggs at any time from signing the informed consent through 1 month after receiving the last dose of the trial V160/placebo.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2200 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (95):
- United States (54):
  - Alabama Clinical Therapeutics ( Site 0025), Birmingham, Alabama
  - Achieve Clinical Research, LLC ( Site 0055), Birmingham, Alabama
  - Synexus US Phoenix Southeast ( Site 0057), Chandler, Arizona
  - Inland Empire Liver Foundation ( Site 0026), Rialto, California
  - Integrated Research of Inland, Inc. ( Site 0042), Riverside, California
  - California Research Foundation ( Site 0286), San Diego, California
  - Bayview Research Group, LLC ( Site 0012), Valley Village, California
  - Diablo Clinical Research, Inc ( Site 0009), Walnut Creek, California
  - Emerson Clinical Research Institute ( Site 0297), Washington D.C., District of Columbia
  - Clinical Research of South Florida ( Site 0047), Coral Gables, Florida
  - Indago Research & Health Center, Inc ( Site 0007), Hialeah, Florida
  - NF Research Center LLC ( Site 0013), Hialeah, Florida
  - Best Quality Research Inc. ( Site 0031), Hialeah, Florida
  - Care Partners Clinical Research, LLC ( Site 0002), Jacksonville, Florida
  - L&C Professional Medical Research Institute ( Site 0021), Miami, Florida
  - Advanced Medical Research Institute ( Site 0296), Miami, Florida
  - Kendall South Medical Center, Inc ( Site 0008), Miami, Florida
  - New Age Medical Research Corporation ( Site 0018), Miami, Florida
  - Clinical Associates of Orlando, LLC ( Site 0032), Orlando, Florida
  - Columbus Regional Research Institute ( Site 0298), Columbus, Georgia
  - Heartland Research Associates, LLC ( Site 0044), Augusta, Kansas
  - Heartland Research Associates, LLC ( Site 0023), Newton, Kansas
  - Heartland Research Associates, LLC ( Site 0019), Wichita, Kansas
  - ACC Pediatric Research ( Site 0022), Haughton, Louisiana
  - University of Maryland School of Medicine ( Site 0041), Baltimore, Maryland
  - St Michaels Med Center ( Site 0285), Newark, New Jersey
  - Albuquerque Clinical Trials ( Site 0052), Albuquerque, New Mexico
  - Mid Hudson Medical Research ( Site 0294), New Windsor, New York
  - Carolina Women's Research and Wellness Center ( Site 0035), Durham, North Carolina
  - PMG Research of Raleigh, LLC ( Site 0048), Raleigh, North Carolina
  - PMG Research of Wilmington ( Site 0006), Wilmington, North Carolina
  - Cincinnati Children's Hospital Medical Center ( Site 0003), Cincinnati, Ohio
  - Senders Pediatrics ( Site 0060), Cleveland, Ohio
  - Rapid Medical Research, Inc. ( Site 0038), Cleveland, Ohio
  - Lynn Health Science Institute ( Site 0287), Oklahoma City, Oklahoma
  - Coastal Pediatric Research ( Site 0010), Charleston, South Carolina
  - Parkside Pediatric ( Site 0288), Greenville, South Carolina
  - Coastal Carolina Research Center ( Site 0053), Mt. Pleasant, South Carolina
  - Palmetto Clinical Research ( Site 0289), Summerville, South Carolina
  - Tekton Research, Inc. ( Site 0036), Austin, Texas
  - Coastal Bend Clinical Research ( Site 0299), Corpus Christi, Texas
  - Radiant Research - Dallas ( Site 0045), Dallas, Texas
  - University of Texas Medical Branch at Galveston ( Site 0049), Galveston, Texas
  - Juno Research, LLC ( Site 0293), Houston, Texas
  - Accurate Clinical Management, LLC ( Site 0028), Pasadena, Texas
  - Diagnostics Research Group ( Site 0001), San Antonio, Texas
  - Synexus Research ( Site 0058), San Antonio, Texas
  - Crossroads Clinical Research LLC ( Site 0283), Victoria, Texas
  - Health Research of Hampton Roads, Inc. ( Site 0014), Newport News, Virginia
  - Clinical Research Associates of Tidewater ( Site 0056), Norfolk, Virginia
  - York Clinical Research, LLC ( Site 0033), Norfolk, Virginia
  - National Clinical Research-Richmond, Inc. ( Site 0051), Richmond, Virginia
  - Multicare / Rockwood Clinic ( Site 0034), Spokane, Washington
  - Premier Clinical Research Group ( Site 0050), Spokane, Washington
- Australia (5):
  - Paratus Clinical Pty Ltd - Blacktown Clinic ( Site 0247), Blacktown, New South Wales
  - Paratus Clinical Kanwal - Trial Clinic ( Site 0243), Kanwal, New South Wales
  - Holdsworth House Medical Practice ( Site 0241), Sydney, New South Wales
  - University of the Sunshine Coast Clinical Trials Centre ( Site 0244), Morayfield, Queensland
  - University of the Sunshine Coast Clinical Trials Centre ( Site 0245), Sippy Downs, Queensland
- Canada (8):
  - Vaccine Evaluation Center ( Site 0264), Vancouver, British Columbia
  - PrimeHealth Clinical Research ( Site 0070), Toronto, Ontario
  - Clinique OVO ( Site 0067), Montreal, Quebec
  - McGill University Health Centre - Vaccine Study Centre ( Site 0064), Pierrefonds, Quebec
  - CHUQ - Unite de Recherche en Sante Publique ( Site 0065), Québec, Quebec
  - Diex Recherche Quebec Inc ( Site 0069), Québec, Quebec
  - Diex Recherche Sherbrooke Inc. ( Site 0066), Sherbrooke, Quebec
  - Diex Recherche Victoriaville Inc. ( Site 0068), Victoriaville, Quebec
- Finland (10):
  - Tampereen yliopisto Espoon rokotetutkimusklinikka ( Site 0186), Espoo
  - Tampereen yliopisto Etela-Helsingin Rokotetutkimusklinikka ( Site 0188), Helsinki
  - Ita-Helsingin Rokotetutkimuskeskus ( Site 0184), Helsinki
  - Jarvenpaan rokotetutkimuskeskus ( Site 0185), Jarvenpaa
  - Tampereen yliopisto Kokkolan rokotetutkimusklinikka ( Site 0190), Kokkola
  - Tampereen yliopisto Oulun rokotetutkimusklinikka ( Site 0187), Oulu
  - Pori Vaccine Research Center ( Site 0182), Pori
  - Seinajoki Vaccine Research Center ( Site 0189), Seinäjoki
  - Tampereen yliopisto Rokotetutkimuskeskus ( Site 0181), Tampere
  - Turku Vaccine Research Center ( Site 0183), Turku
- Israel (8):
  - Rambam Medical Center - Health Care Campus ( Site 0219), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 0216), Jerusalem
  - Meir MC ( Site 0213), Kfar Saba
  - Western Galilee Hospital ( Site 0212), Nahariya
  - Rabin Medical Center ( Site 0218), Petah Tikva
  - Sakhnin west neighbourhood ( Site 0211), Sakhnin
  - Sourasky Medical Center ( Site 0217), Tel Aviv
  - Maccabi Healthcare Services ( Site 0220), Tel Aviv
- Russia (6):
  - Limited Liability Company Medical Centre Aibolit ( Site 0229), Kazan'
  - LLC Scientific Research Medical Complex Your Health. ( Site 0230), Kazan'
  - City Clinical Hospital 13 of Moscow ( Site 0232), Moscow
  - Antenatal clinic #22 ( Site 0225), Saint Petersburg
  - Siberian State Medical University ( Site 0231), Tomsk
  - Central City Hospital 7 ( Site 0237), Yekaterinburg
- Spain (4):
  - Hospital Clinic de Barcelona ( Site 0155), Barcelona
  - Hospital Universitario 12 de Octubre ( Site 0152), Madrid
  - Hospital Universitario La Paz ( Site 0157), Madrid
  - Hospital Clinico Universitario de Santiago ( Site 0151), Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Das R, Blazquez-Gamero D, Bernstein DI, Gantt S, Bautista O, Beck K, Conlon A, Rosenbloom DIS, Wang D, Ritter M, Arnold B, Annunziato P, Russell KL; V160-002 study group. Safety, efficacy, and immunogenicity of a replication-defective human cytomegalovirus vaccine, V160, in cytomegalovirus-seronegative women: a double-blind, randomised, placebo-controlled, phase 2b trial. Lancet Infect Dis. 2023 Dec;23(12):1383-1394. doi: 10.1016/S1473-3099(23)00343-2. Epub 2023 Aug 31. PMID 37660711

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of approximately 2100 participants were planned to be enrolled with 2200 participants actually randomized.
Groups:
- V160 3-Dose Regimen: Participants received V160 vaccination by intramuscular (IM) injection on Day 1, Month 2, and Month 6.
- V160 2-Dose Regimen: Participants received V160 vaccination by IM injection on Day 1 and Month 6 and placebo at Month 2.
- Placebo: Participants received placebo by IM injection on Day 1, Month 2, and Month 6.
Period: Overall Study
Arm/Group | V160 3-Dose Regimen | V160 2-Dose Regimen | Placebo
Started | 733 | 733 | 734
Treatment 1 | 729 | 729 | 733
Treatment 2 | 680 | 680 | 679
Treatment 3 | 614 | 631 | 622
Completed | 614 | 631 | 622
Not Completed | 119 | 102 | 112
Not completed — Withdrawal by Subject | 46 | 46 | 52
Not completed — Adverse Event | 8 | 7 | 0
Not completed — Lost to Follow-up | 41 | 24 | 39
Not completed — Non-compliance with Study Drug | 2 | 2 | 0
Not completed — Physician Decision | 5 | 2 | 3
Not completed — Pregnancy | 10 | 12 | 12
Not completed — Protocol Deviation | 2 | 3 | 3
Not completed — Withdrawal by Parent/Guardian | 1 | 2 | 2
Not completed — Randomized but not treated | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V160 3-Dose Regimen | V160 2-Dose Regimen | Placebo | Total
Number analyzed (Participants) | 733 | 733 | 734 | 2200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.0 (5.0) | 26.1 (4.9) | 25.9 (4.9) | 26.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 733 | 733 | 734 | 2200
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 144 | 145 | 143 | 432
  Not Hispanic or Latino | 588 | 585 | 587 | 1760
  Unknown or Not Reported | 1 | 3 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 4 | 5
  Asian | 6 | 7 | 6 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 47 | 49 | 43 | 139
  White | 657 | 652 | 665 | 1974
  More than one race | 23 | 23 | 16 | 62
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Became Infected With Wild-Type Cytomegalovirus Infection Starting at 4 Weeks Post Last Dose (V160 3-dose Regimen Group and Placebo Group)
Description: Cytomegalovirus infection (CMVi) was defined as the detection of wild-type cytomegalovirus (CMV) (non vaccine type) by polymerase chain reaction in a single saliva or urine sample in a previously CMV-uninfected participant. CMVi cases in the 3-dose regimen and placebo groups were reported and incidence rate (per 100 person-years) calculated based on follow-up time starting at 4 weeks post last dose (Month 7) through approximately Month 24 (or time point to reach required cases for assessment). The percent reduction in CMVi incidence rate in the 3-dose regimen group compared to the placebo group was assessed.
Time Frame: 4 weeks post last vaccination (Month 7) up to ~Month 24
Population: The analysis population included participants who were CMV seronegative at Day 1 and CMV negative by polymerase chain reaction (PCR) for nonvaccine strain virus from post Day 1 through Month 7, had received all 3 injections/vaccinations within the vaccination visit window, and did not have any deviations from protocol deemed to potentially interfere with the evaluation of efficacy or immune response to injection of V160.
Measure: Count of Participants; unit: Participants
Arm/Group | V160 3-Dose Regimen | Placebo
Number analyzed (Participants) | 556 | 543
Participants | 14 | 24
Statistical Analysis 1: Comparison: V160 3-Dose Regimen vs Placebo; Test type: Other — The incidence rate per 100 person years (100 x number of CMVi cases/total person-years to CMVi or end of follow-up) is presented along with 95% confidence interval (CI); Incidence Rate Estimate = 2.9, 95% CI 2-sided [1.6 to 4.9]
Statistical Analysis 2: Comparison: V160 3-Dose Regimen vs Placebo; Test type: Other — The incidence rate per 100 person years (100 x number of CMVi cases/total person-years to CMVi or end of follow-up) is presented along with 95% CI; Incidence Rate Estimate = 5.1, 95% CI 2-sided [3.3 to 7.6]
Statistical Analysis 3: Comparison: V160 3-Dose Regimen vs Placebo; Test type: Other — The statistical criterion for success requires the lower limit of the 95% CI of vaccine efficacy (VE) to be greater than 0%; Vaccine Efficacy = 42.4, 95% CI 2-sided [-13.5 to 71.1]

2. Primary Outcome: Number of Participants With Solicited Injection-site Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. Following vaccination with V160 or placebo, the number of participants with solicited injection-site AEs was assessed. The solicited injection-site AEs assessed were redness/erythema, swelling, and pain.
Time Frame: Up to 5 days after each vaccination
Population: The analysis population included all randomized participants who received at least 1 injection of V160 or placebo, had safety follow-up data, and had been assigned to the treatment arm corresponding to the actual clinical material received.
Measure: Count of Participants; unit: Participants
Arm/Group | V160 3-Dose Regimen | V160 2-Dose Regimen | Placebo
Number analyzed (Participants) | 728 | 729 | 732
Participants | 683 | 668 | 249
Statistical Analysis 1: Comparison: V160 3-Dose Regimen vs Placebo; Test type: Other; Difference in Percent = 59.8, 95% CI 2-sided [55.8 to 63.5]
Statistical Analysis 2: Comparison: V160 2-Dose Regimen vs Placebo; Test type: Other; Difference in Percent = 57.6, 95% CI 2-sided [53.5 to 61.5]

3. Primary Outcome: Number of Participants With Solicited Systemic AEs
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. Following vaccination with V160 or placebo, the number of participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were fatigue, joint pain/arthralgia, muscle pain/myalgia, and headache.
Time Frame: Up to 14 days after each vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | V160 3-Dose Regimen | V160 2-Dose Regimen | Placebo
Number analyzed (Participants) | 728 | 729 | 732
Participants | 621 | 633 | 508
Statistical Analysis 1: Comparison: V160 3-Dose Regimen vs Placebo; Test type: Other; Difference in Percent = 15.9, 95% CI 2-sided [11.7 to 20.1]
Statistical Analysis 2: Comparison: V160 2-Dose Regimen vs Placebo; Test type: Other; Difference in Percent = 17.4, 95% CI 2-sided [13.3 to 21.6]

4. Primary Outcome: Number of Participants With Vaccine-related Serious Adverse Events
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine was determined by the investigator. Following vaccination with V160 or placebo, the number of participants with vaccine-related serious adverse events was assessed.
Time Frame: Up to 14 days after each vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | V160 3-Dose Regimen | V160 2-Dose Regimen | Placebo
Number analyzed (Participants) | 728 | 729 | 732
Participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: V160 3-Dose Regimen vs Placebo; Test type: Other; Difference in Percent = 0.0, 95% CI 2-sided [-0.5 to 0.5]
Statistical Analysis 2: Comparison: V160 2-Dose Regimen vs Placebo; Test type: Other; Difference in Percent = 0.0, 95% CI 2-sided [-0.5 to 0.5]

5. Secondary Outcome: Number of Participants Who Became Infected With Wild-Type CMV Infection Starting at 4 Weeks Post Last Dose (V160 2-dose Regimen Group and Placebo Group)
Description: CMVi is defined as detection of wild-type CMV (non-vaccine type) by polymerase chain reaction in a single saliva or urine sample in a previously CMV-uninfected participant. CMVi cases in the 2-dose regimen and placebo groups were reported and incidence rate (per 100 person-years) calculated based on follow-up time starting at 4 weeks post last dose (Month 7) through approximately Month 24 (or time point to reach required cases for assessment). The percent reduction in CMVi incidence rate in the 2-dose regimen group compared to the placebo group was assessed.
Time Frame: 4 weeks post last vaccination (Month 7) up to ~Month 24
Population: The analysis population included participants who were CMV seronegative at Day 1 and CMV negative by polymerase chain reaction (PCR) for nonvaccine strain virus from post Day 1 through Month 7, had received all 2 injections/vaccinations within the vaccination visit window, and did not have any deviations from protocol deemed to potentially interfere with the evaluation of efficacy or immune response to injection of V160.
Measure: Count of Participants; unit: Participants
Arm/Group | V160 2-Dose Regimen | Placebo
Number analyzed (Participants) | 546 | 543
Participants | 31 | 24
Statistical Analysis 1: Comparison: V160 2-Dose Regimen; Test type: Other — [test comment as in outcome 1, analysis 2]; Incidence Rate Estimate = 6.7, 95% CI 2-sided [4.6 to 9.5]
Statistical Analysis 2: Comparison: Placebo; Test type: Other — [test comment as in outcome 1, analysis 2]; Incidence Rate Estimate = 5.1, 95% CI 2-sided [3.3 to 7.6]
Statistical Analysis 3: Comparison: V160 2-Dose Regimen; Test type: Other — [test comment as in outcome 1, analysis 3]; Vaccine Efficacy = -32.0, 95% CI 2-sided [-135.0 to 25.0]

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events: Up to ~Month 24; Non-serious adverse events: Up to 14 days following any vaccination.
Description: The analysis population for the serious and non-serious adverse events included all randomized participants who received at least 1 injection of V160 or placebo, had safety follow-up data, and had been assigned to the treatment arm corresponding to the actual clinical material received. The all-cause mortality analysis population included all randomized participants.
Groups:
- V160 3-Dose Group: Participants received V160 vaccination by intramuscular (IM) injection on Day 1, Month 2, and Month 6.
- V160 2-Dose Group: Participants received V160 vaccination by IM injection on Day 1 and Month 6 and placebo at Month 2.
- Placebo Group: Participants received placebo by IM injection on Day 1, Month 2, and Month 6.
Arm/Group | V160 3-Dose Group | V160 2-Dose Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/733 | 0/733 | 0/734
Serious Adverse Events (participants affected / at risk) | 22/728 | 29/729 | 26/732
Other Adverse Events (participants affected / at risk) | 697/728 | 700/729 | 557/732
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V160 3-Dose Group (N=728) | V160 2-Dose Group (N=729) | Placebo Group (N=732)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pelvic bone injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic arthropathy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Idiopathic intracranial hypertension (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 6 (6) | 7 (7)
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (2)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V160 3-Dose Group (N=728) | V160 2-Dose Group (N=729) | Placebo Group (N=732)
Nausea (Gastrointestinal disorders) | 45 (50) | 55 (68) | 46 (54)
Fatigue (General disorders) | 457 (1128) | 461 (1077) | 357 (843)
Injection site erythema (General disorders) | 254 (400) | 208 (273) | 30 (39)
Injection site pain (General disorders) | 680 (1943) | 664 (1524) | 239 (374)
Injection site pruritus (General disorders) | 44 (54) | 26 (34) | 4 (5)
Injection site swelling (General disorders) | 248 (404) | 233 (311) | 21 (26)
Pyrexia (General disorders) | 75 (93) | 90 (112) | 27 (42)
Nasopharyngitis (Infections and infestations) | 53 (59) | 53 (56) | 37 (40)
Arthralgia (Musculoskeletal and connective tissue disorders) | 162 (226) | 162 (249) | 76 (121)
Myalgia (Musculoskeletal and connective tissue disorders) | 455 (996) | 424 (818) | 200 (336)
Headache (Nervous system disorders) | 434 (988) | 450 (976) | 368 (795)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 62 (81) | 65 (80) | 69 (80)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the sponsor, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT03486834/Prot_SAP_000.pdf